CLINICAL TRIAL: NCT05039606
Title: Prospective, Multicentric, Randomized Clinical Study of Radiotherapy Combined With Nedaplatin Contrast and Cisplatin for the Treatment of Locally Advanced Head and Neck Squamous Carcinoma
Brief Title: Clinical Study of Radiotherapy Combined With Nedaplatin Contrast and Cisplatin for the Treatment of Locally Advanced Head and Neck Squamous Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guiyang Medical University (Other)
Responsible Party: Principal Investigator, Feng Jing, Head and neck cancer director,chief researcher,clinical professor, Guiyang Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210829
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Squamous Carcinoma
Keywords: Local advanced head and neck squamous carcinoma; Nedaplatin; Adverse reactions; Efficacy
MeSH Terms: interventions — nedaplatin; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the treatment group (Experimental): Nedplatin combined with intensive radiotherapy group
  Interventions: Drug: Nedaplatin
- the control group (Active Comparator): Cisplatin was combined with the IMRT group
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Nedaplatin — Nedaplatin is a second-generation platinum-like derivative, which is a cell cycle non-specific drug, with a mechanism of action and efficacy similar to cisplatin, and a wide anti-cancer spectrum
  Arms: the treatment group
Drug: Cisplatin — Cisplatin, aka cis-dichlorodiamineplatin, is a platinum-containing anticancer drug
  Arms: the control group

SUMMARY:
This study was designed as a prospective, multicenter and randomized clinical study of radiotherapy combined with Nedaplatin contrast and cisplatin for local advanced head and neck squamous SCC, aiming to explore the efficacy, safety and long-term efficacy of this trial and control groups and provide some evidence for the selection of clinical treatment options.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) is a common malignancy accounting for more than 90% of head and neck tumors and over 60% of patients with mid-to late stage (-b) stage at diagnosis.For patients with moderate and advanced head and neck squamous carcinoma, concurrent chemoradiotherapy and chemotherapy is recommended for category 1 and the preferred drug is cisplatin.The application of simultaneous chemoradiotherapy can significantly improve the overall survival rate of patients with locally advanced head and neck squamous carcinoma, and effectively reduce their local recurrence rate and distant metastasis rate.However, the application of cisplatin aggravates the toxic and side reactions, such as nausea and vomiting, radioactive oral mucosal response, nephrotoxicity and ear toxicity.Although the clinical benefit of synchronous chemochemotherapy of locally advanced head and neck squamous carcinoma with cisplatin as chemotherapy is considerable, due to its obvious toxic and side reaction, some patients can not tolerate, cannot complete the whole course of treatment and quality of life, resulting in a substantial reduction in the treatment effect.Therefore, in synchronous chemoradiotherapy of locally advanced head and NSCC, there is an urgent need to find an efficient, hypotoxic, novel chemotherapeutic agent to address this problem.

Nedaplatin is the second generation platinum derivative, for cell cycle nonspecific drugs, mechanism and efficacy similar to cisplatin, anticancer spectrum, and cisplatin without drug resistance, cisplatin resistance still has a good effect, its gastrointestinal reaction and nephrotoxicity is significantly reduced, main dose-limiting toxicity, grade marrow suppression, clinical application without hydration, patients good tolerance and convenient to use, can significantly improve the quality of life of patients.A number of foreign studies have found that nedaplatin combination chemotherapy is effective in esophageal cancer, non-small cell lung cancer and cervical cancer, patients are tolerated, and the digestive tract response is significantly reduced, which helps to ensure the integrity of the course of treatment.Wang Zhennan and other studies reported that nedaplatin can improve the radiosensitivity of NPC CNE-2 cells and show dose-dependent inhibition of tumor cells.Koizumi et al also found that nedaplatin with radiotherapy could effective sensitization.In addition, the results of a phase III randomized controlled trial from the Cancer Center of Sun Yat-sen University, which showed that the overall efficiency of nedaplatin combined radiotherapy for local advanced NPC and 2-year progression-free survival rate were no less than cisplatin (88.7%vs89.7%), and compared with the cisplatin group, gastrointestinal loss, nausea, vomiting and weight loss quality score were significantly improved.

ELIGIBILITY:
Inclusion Criteria:

1. voluntarily participated and signed the informed consent form in writing
2. is 18-70 and gender unlimited
3. histologically proved to be squamous cell carcinoma
4. as AJCC(version 8): -A, ⅣB head and neck squamous carcinoma unable or denied surgery; ~ A, ⅣB squamous carcinoma of the head and neck with the following postoperative risk factors: positive or proximal resection, lymph node envelope invasion, nerve and vascular invasion, primary focal pT3 or T4, N2 or N3 lymph node lesions.
5. card score ≥ 70
6. survival is expected to be ≥ for 6 months
7. fertility women should guarantee contraception during entering the study
8. Hemoglobin (HGB) ≥ 100 g/L, leukocyte (WBC) ≥ 3.5 × 10^9 / L*(unit normal), Platelet (PLT) ≥ 100 × 10^9 / L(unit normal), neutrophil (WBC) ≥ 1.5 × 10^9 / L*(unit normal)
9. liver function: 2.5 times of the upper normal limit (ULN), gluten transaminase (ASAT) <; total bilirubin <1.5 × ULN
10. renal function: Serum creatinine <ULN, endogenous creatinine clearance (Ccr) ≥ 55 ml/min
11. has no severe complications such as hypertension, diabetes, coronary heart disease, and psychiatric history
12. (no history of head and neck radiotherapy or chemotherapy within 3 months)

Exclusion Criteria:

1. has a distant transfer
2. has received epidermal growth factor targeted or immunotherapy
3. has developed other malignant tumors (except for cured basal cell carcinoma or cervical carcinoma in situ)
4. pregnant women or lactating women and women of childbearing age who refuse contraception during the treatment observation period
5. has a serious history of severe allergies or abnormalities
6. refused or cannot sign an informed consent to participate in the trial
7. substance abuse or alcohol addicts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
NCI CTCAE 5.0 | 1 year
  Acute virulence side response
RESIST1.1 | 1year
  Use to assess recent efficacy

SECONDARY OUTCOMES:
overall survival | 5 years
  Overall survival was assessed at 5 years after the end of chemoradiotherapy during the same period
Progression-free survival rate | 5 years
  Progression-free survival rate was assessed at 5 years after the end of chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Feng Jin, Bachelor, Study Chair — The Affiliated Cancer Hospital of Guizhou Medical University
Locations (1):
- The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No